CLINICAL TRIAL: NCT05723562
Title: A Phase 2, Single-Arm, Open-Label Study With Dostarlimab Monotherapy in Participants With Untreated Stage II/III dMMR/MSI-H Locally Advanced Rectal Cancer
Brief Title: A Study of Dostarlimab in Untreated dMMR/MSI-H Locally Advanced Rectal Cancer
Acronym: AZUR-1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219369; 2022-003289-18 (EudraCT Number)
Record Dates: First submitted 2023-02-02; First posted 2023-02-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms, Rectal
Keywords: JEMPERLI; dostarlimab-gxly; GSK4057190; Stage II/III rectal cancer; Neoadjuvant; dMMR; MSI-H
MeSH Terms: conditions — Rectal Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dostarlimab monotherapy (Experimental)
  Interventions: Biological: Dostarlimab

INTERVENTIONS:
Biological: Dostarlimab — Dostarlimab will be administered.
  Other Names: JEMPERLI; dostarlimab-gxly; TSR-042; GSK4057190

SUMMARY:
The purpose of this study is to investigate dostarlimab monotherapy in participants with locally advanced Mismatch-repair deficient (dMMR)/Microsatellite instability-high (MSI-H) rectal cancer who have received no prior treatment. Participants who achieve complete clinical response (cCR) following dostarlimab treatment will undergo non-operative management (NOM), including close surveillance for recurrent disease. The goal of the study is to determine if Dostarlimab therapy alone is an effective treatment that can allow participants to avoid chemotherapy, radiation, and surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically confirmed Stage II to III (T3-T4, N0, or T any, N+), locally advanced rectal cancer
* Participant has radiologically and endoscopically evaluable disease.
* Participant has a tumor which can be categorized as dMMR or MSI-H by local or central assessment

Exclusion Criteria:

* Participant has distant metastatic disease.
* Participant has received prior radiation therapy, systemic therapy, or surgery for management of rectal cancer.
* Participant has any history of interstitial lung disease or pneumonitis
* Participant has experienced any of the following with prior immunotherapy: any imAE of Grade ≥3, immune-related severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (Stevens-Johnson Syndrome, toxic epidermal necrolysis, or DRESS syndrome), or myocarditis of any grade. Non clinically significant laboratory abnormalities are not exclusionary.
* Participant has a known additional malignancy that progressed or required active treatment within the past 2 years. Exceptions include adequately treated superficial skin cancers, superficial bladder cancers, and other in situ cancers.
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Participant has a history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies, fusion proteins, or has known allergies to dostarlimab or its excipients.
* Has received or plans to receive an organ or stem cell transplant that uses donor stem cells (allogeneic stem cell transplant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2029-10-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Sustained Complete Clinical Response for 12 Months (cCR12) as assessed by Independent Central Review (ICR) | 18 Months
  cCR12 is achieved when a participant maintains complete clinical response (cCR) as assessed by ICR for 12 months following their post-intervention disease assessment (PIDA)

SECONDARY OUTCOMES:
Number of Participants with Sustained Complete Clinical Response for 24 Months (cCR24) as assessed by ICR | 30 Months
  cCR24 is achieved when a participant maintains complete clinical response (cCR) as assessed by ICR for 24 months following their post-Intervention disease assessment (PIDA)
Number of Participants with Sustained Complete Clinical Response for 36 Months (cCR36) as assessed by ICR | 42 Months
  cCR36 is achieved when a participant maintains complete clinical response (cCR) as assessed by ICR for 36 months following their post-Intervention disease assessment (PIDA)
Number of Participants with Event Free Survival at 3 years (EFS3) as assessed by Investigator | 3 years
  EFS3 is defined as participants who remained alive and free of disease progression precluding surgery, local recurrence, and distant recurrence at 3 years as assessed by Investigator
Event Free Survival (EFS) as assessed by Investigator | Up to 74 months
  EFS is defined as time from the date of first dose of study intervention to any of the following events: progression of disease that precludes surgery, local recurrence, distant recurrence (all as assessed by the investigator), or death due to any cause
Number of Participants with cCR12 as assessed by Investigator | 18 Months
  cCR12 is achieved when a participant maintains complete clinical response (cCR) as assessed by Investigator for 12 months following their post-intervention disease assessment (PIDA)
Number of Participants with cCR24 as assessed by Investigator | 30 Months
  cCR24 is achieved when a participant maintains complete clinical response (cCR) as assessed by Investigator for 24 months following their post-intervention disease assessment (PIDA)
Number of Participants with cCR36 as assessed by Investigator | 42 Months
  cCR36 is achieved when a participant maintains complete clinical response (cCR) as assessed by Investigator for 36 months following their post-intervention disease assessment (PIDA)
Objective Response Rate (ORR) assessed by ICR | Up to 33 Weeks
  ORR is defined as number of participants achieving a partial response (PR), near complete response (nCR) or complete clinical response (cCR) at PIDA or at least 4 weeks but no longer than 8 weeks after PIDA for participants with nCR or incomplete clinical response (iCR) (PIDA 2) as assessed by ICR
Objective Response Rate (ORR) as assessed by Investigator | Up to 33 Weeks
  ORR by Investigator, defined as achieving a PR, nCR, or cCR at PIDA or at least 4 weeks but no longer than 8 weeks after PIDA for participants with nCR or iCR
Organ Preservation Rate | 3 years
  Organ Preservation Rate defined as not undergoing Total Mesorectal Excision (TME), either as primary management or for local recurrence, and who did not have a permanent colostomy created, at any time up to 3 years
Disease-Specific Survival (DSS) | Up to 74 months
  DSS is defined as time from the date of first dose of study intervention to death due to disease
Disease-Specific Response at 5 years (DSS5) | Up to 5 years
  DSS5 is defined as the number of participants not dying due to disease under study at 5 years from the first dose of study intervention
Overall Survival (OS) | Up to 74 months
  OS is defined as time from first dose of study intervention to death from any cause
Overall Survival at 5 years (OS5) | Up to 5 years
  OS is defined as number of participants as being alive at 5 years from first dose of study intervention
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs), Immune mediated Adverse Events (imAEs) based on Severity | Up to 74 months
Number of Participants with discontinuation of study intervention | Up to 24 weeks
Serum concentration of Dostarlimab | Up to 37 weeks
Concentration at the end of infusion (C-EOI) of Dostarlimab | Up to 37 weeks
Trough Concentration (C-trough) of Dostarlimab | Up to 37 weeks
Number of Participants with Anti-Drug Antibodies against Dostarlimab | Up to 37 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (37):
- United States (7):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richmond, Virginia
- Canada (4):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- France (5):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rennes
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Düsseldorf
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, München
- Italy (3):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Roma
- Japan (3):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
- GSK Investigational Site, Utrecht, Netherlands
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Valencia
- United Kingdom (3):
  - GSK Investigational Site, Leeds West Yorkshire
  - GSK Investigational Site, London
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.